CLINICAL TRIAL: NCT02048904
Title: Clinical Effect of Dipeptidyl Peptidase-4 (DPP-4) Inhibitors in Urinary Albumin to Creatinine Ratio in Patients With Overt Kidney Disease
Brief Title: Use of Sitagliptin to Decrease Microalbuminuria
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Original Principal Investigator left institution. No data analyzed.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1207397
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes; Microalbuminuria
Keywords: microalbuminuria; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Active Comparator): 100 mg/day for 3 months
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): 1 pill/day for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg/day for 3 months
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Placebo — Placebo 1 pill/day for 3 months
  Arms: Placebo

SUMMARY:
The people being asked to participate in this study have type 2 diabetes and abnormal levels of protein in their urine. This indicates that they are starting to develop diabetic kidney disease. The standard treatment for this is the use of one of two blood pressure medicines, either an angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB). However, these medicines are not always completely effective in stopping/reversing the kidney disease. Some studies have previously suggested that another type of medicine, called sitagliptin, normal used to treat diabetes may also help prevent diabetic kidney disease from getting worse.

This study is being performed to test the effectiveness of sitagliptin as compared to a placebo, along with a stable dose of an ACE inhibitor or ARB, to determine whether or not it will reduce protein levels in their urine. Protein levels in the urine are a marker of the severity of kidney disease.

DETAILED DESCRIPTION:
The people being asked to participate in this study have type 2 diabetes and abnormal levels of protein in their urine. This indicates that they are starting to develop diabetic kidney disease. The standard treatment for this is the use of one of two blood pressure medicines, either an ACE inhibitor or ARB. However, these medicines are not always completely effective in stopping/reversing the kidney disease. Some studies have previously suggested that another type of medicine, called sitagliptin, normal used to treat diabetes may also help prevent diabetic kidney disease from getting worse.

ELIGIBILITY:
Inclusion Criteria:

* Albumin/creatinine ratio between 30-299 mg/dl.
* type 2 diabetes mellitus (T2DM) with hemoglobin A1c between 7 and 9%.
* Stable BP control of less than 145/90 on treatment with ACE or ARB for more than three months prior and during the trial.
* Glomerular filtration rate (GFR) of 60 mL/min/1.73m2 or more.
* Age between 18-75 years old.
* For women: at least two years postmenopausal, surgically sterile, or using an acceptable contraceptive regiment to include oral contraceptive pill (OCP), intrauterine device (IUD), double barrier, depo-provera, or subcutaneous progestin implant and negative urine pregnancy test at trial start.

Exclusion Criteria:

* Pregnancy.
* GFR less than 60 mL/min/73m2.
* Have a history of malignancy other than basal cell or squamous cell skin cancer and have not yet been treated, are currently being treated, or were diagnosed less than 5 years prior to Visit 1.
* Advanced liver disease.
* Subjects cannot be on DPP-4 inhibitor or glycolipoprotein (GLP-1) agonist for at least 4 months before the study start.
* Psychiatric condition that would prevent subject from following directions. Per PI discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Lastra Gonzalez, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia: Diabetes Center, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total enrollment at time of termination of study was 142 participants. However, study was terminated during the enrollment period due to difficulties at the study site. All data collected from participants remains untabulated and no analysis is expected.
Pre-assignment Details: 65 participants had completed study by time of study termination.
Groups:
- Sitagliptin or Placebo: 100 mg/day for 3 months or 1 pill/day for 3 months
  Sitagliptin: Sitagliptin 100 mg/day for 3 months or Placebo: Placebo 1 pill/day for 3 months
Period: Overall Study
Arm/Group | Sitagliptin or Placebo
Started | 142
Completed | 65
Not Completed | 77
Not completed — Withdrawal by Subject | 7
Not completed — Physician Decision | 70

BASELINE CHARACTERISTICS:
Population: Total enrollment was 142 participants, with 65 completing, 7 withdrew voluntarily, and 70 were found to be ineligible. However, data was not analyzed and results are unavailable as investigator and study coordinator no longer work at the institution and did not make information available. Study was terminated prematurely.
Arm/Group | Sitagliptin or Placebo
Number analyzed (Participants) | 65
Age, Customized [Count of Participants; unit: Participants] — Population: Total enrollment was 142 participants, with 65 completing. However, data was not analyzed and results are unavailable as investigator and study coordinator no longer work at the institution and did not make information available. Study was terminated prematurely.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Total enrollment was 142 participants, with 65 completing. However, data was not analyzed and results are unavailable as investigator and study coordinator no longer work at the institution and did not make information available. Study was terminated prematurely.

OUTCOME MEASURES:

1. Primary Outcome: Change in Microalbuminuria Level
Description: Decrease in microalbuminuria level
Time Frame: Six months
Population: Zero participants were analyzed due to early termination of study related to technical/operational difficulties at the study site.
Arm/Group | Sitagliptin or Placebo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Sitagliptin or Placebo
All-Cause Mortality (participants affected / at risk) | 0/142
Serious Adverse Events (participants affected / at risk) | 0/142
Other Adverse Events (participants affected / at risk) | 0/142

LIMITATIONS AND CAVEATS:
Study was terminated during the enrollment period due to difficulties at the study site. 65 participants had completed study by time of study termination.No data were collected or analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No